CLINICAL TRIAL: NCT07235891
Title: Investigating the Impact of Finerenone on Retinal Vascular Dysfunction in Patients With Chronic Kidney Disease
Brief Title: Retinal Protective Effects of Novel Finerenone in Patients With Chronic Kidney Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Merna Abou Khatwa, Assistant Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0202162
Record Dates: First submitted 2025-09-16; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Retinal Nerve Fiber Layer Thickness; Chronic Kidney Disease
Keywords: Retinal dysfunction; Finerenone; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Finerenone) (Experimental): Treatment arm: will receive oral Finerenone in addition to standard treatment.
  Initial dose of finerenone will be determined according to eGFR:
  eGFR>= 60 mL/min: 20 mg once daily. eGFR>25 mL/min, <60 mL/min: 10 mg once daily eGFR<15 mL/min: use is contraindicated Maintenance dose will be determined by the serum potassium level measured 4 weeks after initiation of therapy or dose adjustment according to CKD progression
  Interventions: Drug: Finerenone
- Control arm (No Intervention): Control arm: will receive standard treatment according to patient's condition and symptoms.

INTERVENTIONS:
Drug: Finerenone — Finerenone, a novel orally administered selective non-steroidal MRA demonstrates stronger affinity to the mineralocorticoid receptor (MR) in comparison with eplerenone and spironolactone resulting in better efficacy in aldosterone's inhibition.
  Arms: Intervention arm (Finerenone)

SUMMARY:
Interestingly, A hypothesis-generating analysis was conducted from two studies using routine ophthalmological examinations from clinical trial participants (ReFineDR/DeFineDR), suggesting a potential benefit of finerenone in the delay of progression of non-proliferative diabetic retinopathy (NPDR), independent of baseline HbA1c. Potential benefits of finerenone were also observed in the prevention of required ocular interventions. However, the studies relied on routine ophthalmological examinations done retrospectively, which may have affected data quality and certainly affected quantity. Hence, there is a compelling need to conduct randomized studies with adequate power to detect a potential benefit of finerenone in delaying retinopathy progression, particularly given the lack of alternative options for oral treatment of retinopathy.

DETAILED DESCRIPTION:
An Open labelled, prospective, two-arm, parallel group, non-placebo controlled clinical trial to elucidate the difference in field vision and optical coherence tomography (OCT) metrics 1 month, 3 months and 6 months after treatment initiation compared to baseline findings; OCT metrics include macular thickness, retinal thickness, choroidal thickness, macular ganglion cell-inner plexiform layer and retinal nerve fiber layer (RNFL) thickness.

• According to literature, patients with chronic kidney disease have choroidal and retinal thinning compared to matched healthy volunteers, that's why it is interesting to investigate the potential benefit of finerenone on their retinal metrics.

Both study groups (treatment group) and (control group) will undergo ocular examinations (OCT and field of vision) in addition to blood and urine samples to be obtained at baseline, and at different follow up periods (1 month, 3 months and 6 months).

• Delta changes in field vision and optical coherence tomography (OCT) metrics 1 month, 3 months and 6 months after treatment initiation compared to baseline findings and also between groups will be measured.

Additionally,

* Mean change from baseline scores of routine laboratory investigations of CKD patients including serum creatinine, urea, uric acid, urinary Albumin to creatinine ratio (ACR).
* Mean change from baseline values of metabolic parameters including random blood glucose (RBG), glycated hemoglobin (HbA1C), lipid profile and liver enzymes (ALT and AST). In addition to mean change in body weight.
* To examine the metabolic regulatory effects exhibited by finerenone by measuring the mean change from baseline levels of adipokine leptin.

ELIGIBILITY:
Inclusion Criteria:

* Age: above 18 years
* Diabetic and non-diabetic non-hemodialysis CKD patients (Stage 2 - Stage 4).

Exclusion Criteria:

* Patients on hemodialysis (HD).
* Serum potassium level > 5.5 mEq/L
* Prior/planned ocular interventions (retinal laser treatment, intravitreal injection or vitrectomy).
* Pregnant and lactating women
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Retinal protection | 6 months
  To elucidate the difference in retinal nerve fiber layer (RNFL) thickness (measured in micro meters) measured by optical coherence tomography (OCT) after treatment initiation compared to baseline findings measured by the same device and assessed by the same operator.

SECONDARY OUTCOMES:
CKD progression | 6 months
  Mean change from baseline scores of full renal profile of CKD patients including serum creatinine (mg/dL), urea (mg/dL), uric acid (mg/dL), urinary albumin to creatinine ratio (ACR) (mg/g) and serum albumin (g/dL).
Safety assessment (Number of patients with adverse events) | 6 months
  Safety will be assessed at all scheduled visits by measuring the serum potassium level. Hyperkalemia is an adverse event of special interest in this study. Serum potassium (mmol/L) and hyperkalemia will be characterized through monitoring the change from baseline in serum potassium and identification of the number of patients with serum potassium levels >5.5 mmol/L and >6.0 mmol/L.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-05-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT07235891/Prot_000.pdf